CLINICAL TRIAL: NCT05867940
Title: Effects of Physical Activity on Prescription (PAP) as an Individualised and Health-enhancing Intervention for Children, Adolescents and Adults With Different Disabilities Including Health Economic Analysis
Brief Title: Effects of Physical Activity on Prescription (PAP) as a Health-enhancing Intervention in People With Disabilities
Acronym: PAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dnr 2022-03514-01
Record Dates: First submitted 2023-05-02; First posted 2023-05-22 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Physical Inactivity; Cerebral Palsy; Autism; Autism Spectrum Disorder; Intellectual Disability; Disability Physical; Sedentary Behavior
Keywords: Physical activity on prescription; Children; Adolescents; Adults; Individualised intervention; Participation; Health-enhancing physical activity; Disabilities; Physical disability; Intellectual disability; Autism; Cerebral palsy
MeSH Terms: conditions — Sedentary Behavior; Cerebral Palsy; Autistic Disorder; Autism Spectrum Disorder; Intellectual Disability

STUDY DESIGN:
Intervention Model Description: Four groups of participants will be included in this study; 1) children and adolescents with physical disabilities, 2) children and adolescents with intellectual disabilities, 3) children and adolescents with autism, and 4) adults with physical or intellectual disabilities, or with autism.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Children and adolescents with physical disabilities (Active Comparator): 20 children and adolescents with physical disabilities will participate in physical activity on prescription (PAP). They will be their own controls and will be compared with the other groups. Therefore, there is a baseline 1 and a baseline 2, with 3 months inbetween. After baseline 2, each participant will perform their PAP during 3 months. Assessments to evaluate the results will be performed directly after the 3 months PAP period, and after 6, 12 and 24 months.
  Interventions: Behavioral: Physical activity on prescription
- Children and adolescents with intellectual disabilities (Active Comparator): 20 children and adolescents with intellectual disabilities will participate in physical activity on prescription (PAP). They will be their own controls and will be compared with the other groups. Therefore, there is a baseline 1 and a baseline 2, with 3 months inbetween. After baseline 2, each participant will perform their PAP during 3 months. Assessments to evaluate the results will be performed directly after the 3 months PAP period, and after 6, 12 and 24 months.
  Interventions: Behavioral: Physical activity on prescription
- Children and adolescents with autism (Active Comparator): 20 children and adolescents with autism will participate in physical activity on prescription (PAP). They will be their own controls and will be compared with the other groups. Therefore, there is a baseline 1 and a baseline 2, with 3 months inbetween. After baseline 2, each participant will perform their PAP during 3 months. Assessments to evaluate the results will be performed directly after the 3 months PAP period, and after 6, 12 and 24 months.
  Interventions: Behavioral: Physical activity on prescription
- Adults with physical or intellectual disabilities, or with autism (Active Comparator): 20 adults with physical or intellectual disabilities, or with autism will participate in physical activity on prescription (PAP). They will be their own controls and will be compared with the other groups. Therefore, there is a baseline 1 and a baseline 2, with 3 months inbetween. After baseline 2, each participant will perform their PAP during 3 months. Assessments to evaluate the results will be performed directly after the 3 months PAP period, and after 6, 12 and 24 months.
  Interventions: Behavioral: Physical activity on prescription

INTERVENTIONS:
Behavioral: Physical activity on prescription — Physical activity on prescription (PAP) is a well-established method to enhance physical activity in adults in primary care. The prescribed activity should lead to moderate increase of the pulse, such as walking, cycling, swimming, or gardening, and should be performed over a longer period of time in order to achieve a change towards a more active lifestyle. The activity may be prescribed by a physiotherapist, physician, nurse, or other health professional. PAP has shown to be feasible to increase participation in physical activity and to reduce sedentary behaviour in children with cerebral palsy.
  Motivational interviewing is used for our PAP with participants with disabilities. During PAP-period, the participants are asked to fill in an activity logbook.
  Other Names: PAP

SUMMARY:
Physical inactivity is an increasing problem in the general population in society. However, in people with disabilities, inactivity is even more frequently reported. Physical activity on prescription (PAP) is a well-established method to enhance physical activity. The prescribed physical activity can be activities such as walking, cycling, swimming, or gardening, and should be performed over a longer period. In children with cerebral palsy, PAP has shown to be feasible to increase participation in physical activity and to reduce sedentary behaviour, and the habilitation services in the Region of Skåne have decided to offer PAP to all children and youth with disabilities. It is of great importance to study these interventions when applied on a broader group of patients than previously studied.

The aim is to study the effects of an individualised and health-enhancing intervention in physically inactive people with autism, intellectual and physical disabilities. Also, the cost-effectiveness of PAP will be studied.

60 physically inactive children, aged 8- 17 years, and 20 adults, with autism, intellectual or physical disability will be included. The participants are recruited by their clinical physiotherapists, who also will be carrying out the PAP-intervention. The self-selected physical activity/activities may either be a physical activity organized by a club and/or an everyday activity such as walking a dog or riding a bicycle to school. Each participant fills in an activity logbook. Motivational interviewing will be used to support the participants. The Canadian Occupational Performance Measure can be used to identify what activities the participants are motivated to do, and to detect changes in the participants' perception of their performance of the activity. Quality of life will be monitored. Physical activity will be measured through the International Physical Activity Questionnaire (IPAQ) and a movement monitor (accelerometer). Study specific questionnaires will be filled in regarding costs and background information. Data on health care use of the participants will retrospectively be collected and studied using the health care database in Region Skåne. Data will be collected at 3 months prior to the intervention, just before the intervention starts, when the intervention is finished, and at 6, 12 and 24 months after the intervention. The study has been approved by the Swedish Ethical Review Authority.

DETAILED DESCRIPTION:
Introduction:

Physical inactivity is an increasing problem in the general population in society. However, in people with disabilities, inactivity is even more frequently reported. Physical activity on prescription (PAP) is a well-established method to enhance physical activity in adults in primary care. The prescribed physical activity should lead to moderate increase of the pulse, such as walking, cycling, swimming, or gardening, and should be performed over a longer period in order to achieve a change towards a more active lifestyle. The activity may be prescribed by a physiotherapist, physician, nurse, or other health professional. In children with cerebral palsy, PAP has shown to be feasible to increase participation in physical activity and to reduce sedentary behaviour, and the habilitation services in the Region of Skåne have decided to offer PAP as an activity-enhancing intervention to all children and youth with disabilities. It is of great importance to study these interventions when applied on a broader group of patients (diagnoses and ages) than previously studied.

Aim:

The aim is to study feasibility as well as health effects of an individualised and health-enhancing intervention in physically inactive people with autism, intellectual or physical disabilities in the Department of Habilitation in the Region of Skåne. Also, cost-effectiveness of the intervention PAP will be studied using health-economic analysis methods.

Material:

In total 60 children, aged 8- 17 years; 20 physically inactive children in each group with autism, intellectual and physical disability will be included. Also, 20 physically inactive adults, aged 18 years and older, with any of the disabilities mentioned above, will be recruited for this intervention study.

Method:

Participants are recruited to this study by their clinical physiotherapists, who also will be carrying out the intervention with their patient in ordinary praxis. The selected activity should be adapted to the individual's interests, functional limitations and resources, and may either be a physical activity organized by a club and/or an everyday activity such as walking a dog or riding a bicycle to school. Each participant should report the dates and length of all activities during the 12 weeks that the study will last in an activity logbook.

Measures:

* Motivational interviewing will be used to support the health enhancing change in lifestyle that PAP is expected to contribute to.
* The participants will be questioned about the amount of physical activity using the International Physical Activity Questionnaire (IPAQ) and will be using an accelerometer to objectively measure the activity during a full week (7 days).
* The Canadian Occupational Performance Measure (COPM) can be used to identify what activities the participants are motivated to do, and to detect changes in the participants perception of his/her performance of the activity.
* The Goal Attainment Scaling (GAS) is used for goal setting. GAS is an individualized outcome measure involving goal selection and goal scaling that is standardized in order to calculate the extent to which a patient's goals are met.
* The participants' perception of health-related quality of life will be monitored using the EuroQol Five-Dimensional Questionnaire, Youth Version (EQ-5D-Y) or EuroQol Five-Dimensional Questionnaire, five-level version for adults (EQ-5D-5L).
* To analyze the costs of the intervention, participants themselves and/or parents will be asked to report level of education, occupation, income, family constitution as well as direct or indirect costs for the selected activity. Also, the physiotherapists will report the amount of hours spent to prepare and carry out the activity as well as evaluate/measure the outcome of the intervention for each participant.

The questionnaires directed to participants and/or parents on background information, health-related quality of life, reports of costs associated with the activity and evaluation will be distributed digitally via e-mail to a secure data capturing system using a unique code for each participant. For COPM, accelerometer and IPAQ data, the physiotherapist will report the results digitally to the secure data capturing system for his/her patient using the unique code for each participant.

The cost- effectiveness will be studied by identifying, measuring, evaluating, and comparing the costs and effects for different interventions. In this project, PAP in people with different disabilities will be compared to a three- month period prior to the PAP intervention started, the participants are their own controls. This means that the comparison option is standard care, which would be the care the participant would have had if/when the intervention was not introduced/started.

Data on health care use of the participants will retrospectively be collected and studied using the health care database in Region Skåne.

Data will be collected at 3 months prior to the intervention, just before the intervention starts, when the intervention is finished, and at 6, 12 and 24 months after the intervention.

Ethics:

The study has been reviewed and approved by the Swedish Ethical Review Authority (Dnr 2022-03514-01).

ELIGIBILITY:
Inclusion Criteria:

* Physical inactivity
* Not meeting the physical activity recommendations
* Much sedentary time
* Physical disability
* Intellectual disability
* Autism
* Living in the Skåne Region in Sweden
* Receiving treatment from the habilitation Services in the Skåne Region, Sweden

Exclusion Criteria:

* Meeting the physical activity recommendations

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-06-05 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Subjective measurement of physical activity | 24 months
  Subjective measurement of physical activity by the IPAQ (international physical activity questionnaire). The IPAQ assesses physical activity over the previous week and asks how long and how frequently individuals participate in walking, moderate-intensity activity, and vigorous-intensity activity.
Objective measurement of physical activity | 24 months
  Measurement of physical activity measured by an accelerometer. The participants will be asked to wear an accelerometer for 7 days at each assessment (baseline 1 and 2, after the intervention, after 6, 12 and 24 months).

SECONDARY OUTCOMES:
Measurement of quality of life | 24 months
  Quality of life measured using the EuroQol Five-Dimensional Questionnaire, Youth Version (EQ-5D-Y) or EuroQol Five-Dimensional Questionnaire, five-level version for adults (EQ-5D-5L)
Functional goal attainment | 24 months
  Each participant's goals will be evaluated through the Goal Attainment Scale. The goal/goals are part of the physical activity prescription. The Goal Attainment Scale is described as an individualized outcome measure involving goal selection and goal scaling that is standardized in order to calculate the extent to which a patient's goals are met.
  GAS comprises of goals divided into a 5-point scale from -2 to +2.
  Current state, before the intervention starts = -2; Achievement of somewhat less than expected goal = -1; Achievement of goal = 0; Achieved somewhat more than expected outcome = +1; Achievement of much more than expected goal = +2
Costs for the family | 24 months
  To analyze the costs of PAP, participants themselves and/or parents will be asked to report direct or indirect costs for the selected activity in a study-specific questionnaire.
Costs for the physiotherapists | 24 months
  The physiotherapists will report the amount of hours spent to prepare and carry out the activity as well as evaluate/measure the outcome of the intervention for each participant in a study specific questionnaire.
Assessment of health care use | 24 months
  Data on health care use of the participants will retrospectively be collected and studied using the health care database in Region Skåne.

CONTACTS AND LOCATIONS:
Overall Officials: Katarina Lauruschkus, PhD, Principal Investigator — Region Skåne Sweden
Locations (1):
- Department of habilitation, Region Skåne, Sweden, Malmo, Sweden